CLINICAL TRIAL: NCT04978610
Title: Virtual Acceptance Commitment Therapy (ACT): A Randomized Controlled Trial to Evaluate a Web-Based Intervention for Stress in Adolescents With Chronic Conditions
Brief Title: Virtual ACT for Adolescent Stress
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of lab resources
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey I Gold, PhD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-20-00665
Record Dates: First submitted 2021-07-07; First posted 2021-07-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Chronic Illness
Keywords: Virtual Therapy; Group Therapy; Chronic Medical Condition; Adolescent
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: After informed consent and assent have been obtained and the patient has successfully met the screening criteria, the patient will be enrolled. The study will commence upon the enrollment of approximately 20 participants, at which point participants will be randomized into the Virtual ACT or waitlist (control) group. The intervention group will begin vACT immediately, while the waitlist receive no intervention during the same 6-week time frame. Both groups will take the same baseline questionnaires and post-questionnaires (post, 1 month, and 3 month). After the vACT intervention group finishes, another 6-week vACT session will be offered to the waitlist. The waitlist group will fill out a post-therapy questionnaire again after their 6-weeks. The parents of both groups will fill out a baseline questionnaire and post questionnaires.
  The investigators will repeat this protocol until 144 participants or 72 caregiver-child dyads.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Immediate) (Experimental): Participants in the intervention group will begin their 6-week vACT sessions first and complete baseline, the weekly surveys during intervention, post, one month follow-up, and three month follow-up.
  Interventions: Behavioral: Virtual Acceptance Commitment Therapy
- Control (Waitlist) (Other): Upon the intervention group's completion of the 6-week long vACT, the control group will then enroll into their own 6-week long ACT intervention. The research protocol for the second 6-week long ACT intervention will mirror the protocol with the original 6-week long ACT intervention, except for one change: participants will NOT complete an additional baseline questionnaire prior to starting the 6-week ACT therapy group. The rest of the protocol remains the same. Namely, before each session, each participant will be required to fill out a short survey on their stress and pain throughout previous week. At the conclusion of the final session, participants will follow the complete post-intervention battery of surveys, which mirrors the baseline measures plus the inclusion of satisfaction surveys assessing the effectiveness of the virtual therapy intervention. Participants will complete the post-intervention follow up battery of questionnaires at 1 and 3 months post-intervention.
  Interventions: Behavioral: Virtual Acceptance Commitment Therapy

INTERVENTIONS:
Behavioral: Virtual Acceptance Commitment Therapy — For a period of 6 continuous weeks, participants will meet weekly in a virtual group ACT session with a licensed psychologist hosted on a secure, HIPAA compliant, Zoom account. Each session is 1.5 hours will focus on one ACT concept including Acceptance, Values, Mindfulness, Cognitive Defusion, Experiential Avoidance, and Willingness and Committed Action. Subjects will be given the opportunity to share their thoughts as well as their responses to the exercises at various points throughout the sessions.
  At the beginning of each session, each participant will be required to fill out a short survey on their stress and pain the preceding week. Participants in the control group will not complete weekly measures. All measures will be completed online via a REDCap survey web link. Follow up measures will mirror initial baseline measures in order to measure the within group and between group changes in study outcomes.

SUMMARY:
This study aims to test the effectiveness of a 6-week long virtual Acceptance Commitment group therapy as a non-pharmaceutical intervention to improving other functional outcomes for adolescents with a chronic medical condition in comparison to no treatment.

DETAILED DESCRIPTION:
Upwards of 40% of children and adolescents/young adults (AYAs) in the United States suffer from at least one chronic medical condition, excluding obesity. The emotional and psychological burden of having a chronic condition in youth can lead this population to experience higher rates of stress, depression, and anxiety in addition to reduced health-related quality of life compared to their healthy peers. Acceptance and Commitment Therapy (ACT) is an intervention that teaches skills such as psychological flexibility, mindfulness, and cognitive defusion that has been shown to significantly improve psychological outcomes and quality of life among children and AYAs with chronic conditions. Few studies, however, have examined the efficacy of this intervention in reducing stress among children and AYAs with chronic conditions delivered in a group, web-based format. The need for virtually administered psychological interventions is especially salient amidst the Covid-19 pandemic as CDC guidelines discourage in-person gatherings and close contact with others. The current study aims to: 1) Determine if a web-based group ACT intervention of 6 sessions is more effective than no intervention (waitlist control) in reducing stress among children and AYAs with chronic conditions, 2) Determine if a web-based group ACT intervention of 6 sessions is more effective than no intervention in improving other functional outcomes among children and AYAs with chronic conditions, 3) Evaluate if a web-based group ACT intervention of 6 sessions improves participants skills in psychological flexibility, mindfulness, and cognitive defusion. Study population: Children and Adolescents/Young Adults (ages 14-21) diagnosed with a chronic medical condition seeking care at Children's Hospital Los Angeles, who are in the normal range of development and are eligible to participate in the study. Study Methodology: The study is a non-blinded, randomized, controlled trial designed to examine the effect of a web-based group ACT intervention on stress, depression, anxiety, health-related quality of life, and adaptive psychological skills in children and AYAs with chronic conditions. Statistical analysis: The primary analysis will involve a two independent samples t-test to compare the mean 6-week PSS scores between the two treatment groups. Secondary analyses will compare treatment groups on other study outcomes.

ELIGIBILITY:
Inclusion Criteria for Children:

1. Children who are English speaking
2. Children who are diagnosed with a chronic illness: Defined as a condition that lasts 1 year or more and requires ongoing medical attention or limits activities of daily living or both (excluding obesity).
3. Children with access to a device with internet and webcam capabilities
4. Children with access to a private setting to participate in the intervention

Inclusion criteria for caregivers:

1. Must be 18 years or older and legal guardian of enrolled child
2. English or Spanish speaking, with an ability to read in their language

Exclusion criteria for children:

1. Known developmental delay that precludes the ability to complete questionnaires or participate in group therapy

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess Change via the Perceived Stress Scale (PSS) | baseline at the start of study, through study competition (up to 6 weeks), change from baseline at 6 weeks, change from baseline at 10 weeks, change from baseline at 18 weeks
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. SS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items and then summing across all scale items with higher scores correlating to more stress. There are ten items total with the minimum value set at 0 and maximum 40 with higher scores correlating to more perceived stress.

SECONDARY OUTCOMES:
Assess Change via the Faces Pain Scale-Revised (FPS-R) | baseline at the start of study, through study competition (up to 6 weeks), change from baseline at 6 weeks, change from baseline at 10 weeks, change from baseline at 18 weeks
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how the patients are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.
Assess Change via the Behavior Assessment System for Children, Third Edition (BASC-3) | baseline at the start of study and change from baseline at 6 weeks
  Parent Rating Scales (PRS) will be used to asses the child's behaviors and emotions. Parents evaluate 173 items on a never, sometimes, often, almost always scale. This is scored using a computer software purchased through Pearson. The raw score is converted to a T-score based on age and gender. The T-score has a mean of 50 and standard deviation of 10. T-scores above 65 are clinically significant in that domain.
Assess Change via the Patient-Reported Outcomes Measurement Information System Pediatric Profile-25 v2.0 (PROMIS-25) | baseline at the start of study, change from baseline at 6 weeks, change from baseline at 10 weeks, change from baseline at 18 weeks
  PROMIS-25 measures quality of life (i.e., depression, anxiety, and pain interference). The 25 items are on a 1-5 scale and are scored using the HealthMeasures Scoring Service with higher scores indicating a lower quality of life.
Assess Change via the Comprehensive Adolescent Severity Inventory (CASI) | baseline at the start of study, change from baseline at 6 weeks, change from baseline at 10 weeks, change from baseline at 18 weeks
  This 18-item measure utilizes a three-point Likert scale (none (1), some (2), a lot (3)) to assess how negatively patients view anxiety symptoms. Items are summed with a higher score indicating greater anxiety sensitivity.
Assess Change via the Acceptance and Action Questionnaire (AAQ-II) | baseline at the start of study and change from baseline at 6 weeks
  This 4-item measure uses 0-4 scale (0 = Not at All True; 4 = Very True) with lower sores correlating with higher psychological flexibility.
Assess Change via Avoidance and Fusion Questionnaire Youth (AFQ-Y) | baseline at the start of study and change from baseline at 6 weeks
  This 4-item measure uses 0-4 scale (0 = Not at All True; 4 = Very True) with higher sores correlating with higher psychological inflexibility.
Assess Change via the Child and Adolescent Mindfulness Measure (CAMM) | baseline at the start of study and change from baseline at 6 weeks
  This 10-item measure uses a 0-4 scale (0 = Not at All True; 4 = Very True) with lower scores correlating to greater mindfulness practices.
Assess Change via the Brief Experiential Avoidance Questionnaire (BEAQ) | baseline at the start of study and change from baseline at 6 weeks
  15-item measure uses a 1-6 scale (1= strongly disagree; 6 = strongly agree) with higher scores associated with higher levels of avoidance and psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gold, PhD, Principal Investigator — Children's Hospital Los Angeles; Nicole Mahrer, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai G, Herten MH, Landgraf JM, Korfage IJ, Raat H. Childhood chronic conditions and health-related quality of life: Findings from a large population-based study. PLoS One. 2017 Jun 2;12(6):e0178539. doi: 10.1371/journal.pone.0178539. eCollection 2017. PMID 28575026
- [Background] Bethell CD, Kogan MD, Strickland BB, Schor EL, Robertson J, Newacheck PW. A national and state profile of leading health problems and health care quality for US children: key insurance disparities and across-state variations. Acad Pediatr. 2011 May-Jun;11(3 Suppl):S22-33. doi: 10.1016/j.acap.2010.08.011. PMID 21570014
- [Background] Buhrman M, Skoglund A, Husell J, Bergstrom K, Gordh T, Hursti T, Bendelin N, Furmark T, Andersson G. Guided internet-delivered acceptance and commitment therapy for chronic pain patients: a randomized controlled trial. Behav Res Ther. 2013 Jun;51(6):307-15. doi: 10.1016/j.brat.2013.02.010. Epub 2013 Mar 14. PMID 23548250
- [Background] Cheng C, Brown RC, Cohen LL, Venugopalan J, Stokes TH, Wang MD. iACT--an interactive mHealth monitoring system to enhance psychotherapy for adolescents with sickle cell disease. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:2279-82. doi: 10.1109/EMBC.2013.6609992. PMID 24110179
- [Background] Compas BE, Jaser SS, Dunn MJ, Rodriguez EM. Coping with chronic illness in childhood and adolescence. Annu Rev Clin Psychol. 2012;8:455-80. doi: 10.1146/annurev-clinpsy-032511-143108. Epub 2011 Dec 20. PMID 22224836
- [Background] Fletcher, L., & Hayes, S. C. (2005). Relational frame theory, acceptance and commitment therapy, and a functional analytic definition of mindfulness. Journal of rational-emotive and cognitive-behavior therapy, 23(4), 315-336.
- [Background] Barnes-Holmes Y, Hayes SC, Barnes-Holmes D, Roche B. Relational frame theory: a post-Skinnerian account of human language and cognition. Adv Child Dev Behav. 2001;28:101-38. doi: 10.1016/s0065-2407(02)80063-5. No abstract available. PMID 11605362
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hoffmann D, Rask CU, Hedman-Lagerlof E, Jensen JS, Frostholm L. Efficacy of internet-delivered acceptance and commitment therapy for severe health anxiety: results from a randomized, controlled trial. Psychol Med. 2021 Nov;51(15):2685-2695. doi: 10.1017/S0033291720001312. Epub 2020 May 14. PMID 32404226
- [Background] Hysing M, Elgen I, Gillberg C, Lie SA, Lundervold AJ. Chronic physical illness and mental health in children. Results from a large-scale population study. J Child Psychol Psychiatry. 2007 Aug;48(8):785-92. doi: 10.1111/j.1469-7610.2007.01755.x. PMID 17683450
- [Background] Lappalainen P, Langrial S, Oinas-Kukkonen H, Tolvanen A, Lappalainen R. Web-based acceptance and commitment therapy for depressive symptoms with minimal support: a randomized controlled trial. Behav Modif. 2015 Nov;39(6):805-34. doi: 10.1177/0145445515598142. Epub 2015 Aug 6. PMID 26253644
- [Background] Moazzezi M, Ataie Moghanloo V, Ataie Moghanloo R, Pishvaei M. Impact of Acceptance and Commitment Therapy on Perceived Stress and Special Health Self-Efficacy in Seven to Fifteen-Year-Old Children With Diabetes Mellitus. Iran J Psychiatry Behav Sci. 2015 Jun;9(2):956. doi: 10.17795/ijpbs956. Epub 2015 Jun 1. PMID 26288639
- [Background] Ataie Moghanloo V, Ataie Moghanloo R, Moazezi M. Effectiveness of Acceptance and Commitment Therapy for Depression, Psychological Well-Being and Feeling of Guilt in 7 - 15 Years Old Diabetic Children. Iran J Pediatr. 2015 Aug;25(4):e2436. doi: 10.5812/ijp.2436. Epub 2015 Aug 24. PMID 26396702
- [Background] Pinquart M, Shen Y. Behavior problems in children and adolescents with chronic physical illness: a meta-analysis. J Pediatr Psychol. 2011 Oct;36(9):1003-16. doi: 10.1093/jpepsy/jsr042. Epub 2011 Aug 1. PMID 21810623
- [Background] Rickardsson J, Zetterqvist V, Gentili C, Andersson E, Holmstrom L, Lekander M, Persson M, Persson J, Ljotsson B, Wicksell RK. Internet-delivered acceptance and commitment therapy (iACT) for chronic pain-feasibility and preliminary effects in clinical and self-referred patients. Mhealth. 2020 Jul 5;6:27. doi: 10.21037/mhealth.2020.02.02. eCollection 2020. PMID 32632365
- [Background] Rodriguez EM, Dunn MJ, Zuckerman T, Vannatta K, Gerhardt CA, Compas BE. Cancer-related sources of stress for children with cancer and their parents. J Pediatr Psychol. 2012 Mar;37(2):185-97. doi: 10.1093/jpepsy/jsr054. Epub 2011 Aug 13. PMID 21841187
- [Background] Sansom-Daly UM, Peate M, Wakefield CE, Bryant RA, Cohn RJ. A systematic review of psychological interventions for adolescents and young adults living with chronic illness. Health Psychol. 2012 May;31(3):380-93. doi: 10.1037/a0025977. Epub 2011 Nov 7. PMID 22059621
- [Background] Sawyer MG, Reynolds KE, Couper JJ, French DJ, Kennedy D, Martin J, Staugas R, Ziaian T, Baghurst PA. Health-related quality of life of children and adolescents with chronic illness--a two year prospective study. Qual Life Res. 2004 Sep;13(7):1309-19. doi: 10.1023/B:QURE.0000037489.41344.b2. PMID 15473509
- [Background] Scott W, Chilcot J, Guildford B, Daly-Eichenhardt A, McCracken LM. Feasibility randomized-controlled trial of online Acceptance and Commitment Therapy for patients with complex chronic pain in the United Kingdom. Eur J Pain. 2018 Apr 28. doi: 10.1002/ejp.1236. Online ahead of print. PMID 29704880
- [Background] Trompetter HR, Bohlmeijer ET, Veehof MM, Schreurs KM. Internet-based guided self-help intervention for chronic pain based on Acceptance and Commitment Therapy: a randomized controlled trial. J Behav Med. 2015 Feb;38(1):66-80. doi: 10.1007/s10865-014-9579-0. Epub 2014 Jun 13. PMID 24923259
- [Background] Varni JW, Limbers CA, Burwinkle TM. Impaired health-related quality of life in children and adolescents with chronic conditions: a comparative analysis of 10 disease clusters and 33 disease categories/severities utilizing the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jul 16;5:43. doi: 10.1186/1477-7525-5-43. PMID 17634123
- [Background] Waters E, Davis E, Nicolas C, Wake M, Lo SK. The impact of childhood conditions and concurrent morbidities on child health and well-being. Child Care Health Dev. 2008 Jul;34(4):418-29. doi: 10.1111/j.1365-2214.2008.00825.x. PMID 19154551
- [Background] Wicksell RK, Melin L, Lekander M, Olsson GL. Evaluating the effectiveness of exposure and acceptance strategies to improve functioning and quality of life in longstanding pediatric pain--a randomized controlled trial. Pain. 2009 Feb;141(3):248-257. doi: 10.1016/j.pain.2008.11.006. Epub 2008 Dec 23. PMID 19108951
- [Background] Wicksell RK, Olsson GL, Hayes SC. Mediators of change in acceptance and commitment therapy for pediatric chronic pain. Pain. 2011 Dec;152(12):2792-2801. doi: 10.1016/j.pain.2011.09.003. Epub 2011 Oct 11. PMID 21995881
- [Background] Witlox M, Kraaij V, Garnefski N, de Waal MWM, Smit F, Hoencamp E, Gussekloo J, Bohlmeijer ET, Spinhoven P. An Internet-based Acceptance and Commitment Therapy intervention for older adults with anxiety complaints: study protocol for a cluster randomized controlled trial. Trials. 2018 Sep 17;19(1):502. doi: 10.1186/s13063-018-2731-3. PMID 30223873
- [Background] Woidneck MR, Morrison KL, Twohig MP. Acceptance and Commitment Therapy for the Treatment of Posttraumatic Stress Among Adolescents. Behav Modif. 2014 Jul;38(4):451-76. doi: 10.1177/0145445513510527. Epub 2013 Nov 20. PMID 24265271